CLINICAL TRIAL: NCT06438016
Title: Exploring the Efficiency of Stress Management Training Programs in Reducing Stress Levels Within Nursing Professionals in a Tertiary Care Center in Nepal
Brief Title: Stress Management Training for Nursing Professionals in a Tertiary Care Center in Nepal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dhulikhel Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Makaju Shrestha, Psychologist, Dhulikhel Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205/2024
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Mental Health
Keywords: Stress; Stress Management; Nursing; Nepal
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Treatment group will obtain stress management whilst the control will not. The control group will obtain stress management one month upon study completion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Management Group (Experimental): Participants in this group will be provided with a demographic questionnaire, the DASS-21 and the PSS one week prior to and after the stress management training. The treatment group will be sub-divided into 2 groups of 20-25 participants and subjected to a 4-session stress management training program over the course of 4-weeks (one 40 minute session each week). The DASS and the PSS will be administered to this group one week and one month post completion of the final stress management training session.
  Interventions: Behavioral: Stress Management Training
- Control Group (No Intervention): This control group will fill out the DASS-21 and PSS with the treatment group prior to the treatment group commencing stress management and will also fill out the DASS-21 and PSS upon completion of the treatment group's stress management training. This group will however not obtain stress management training during the study. Training will be provided upon study completion.

INTERVENTIONS:
Behavioral: Stress Management Training — The intervention will comprise of 4 sessions delivered over 4 weeks. The training session will be structured as follows: Session 1 - Psychoeducation relating to stress and its effects. Session 2 - Behavioral techniques to cope with stress 1, Session 3 - Cognitive techniques to cope with stress and Session 4- Behavioral techniques to cope with stress. Both verbal and written means will be used to provide this training.
  Arms: Stress Management Group

SUMMARY:
The goal of this clinical trial is to learn if stress management programs can help alleviate existing and prevent future symptoms of stress in nursing professionals working in a tertiary care center in Nepal.

Researchers will compare the treatment group (exposed to stress management training) to the control group (not exposed to stress management training) to see if

1. Stress management sessions lead to reduction of levels of stress among nurses at tertiary level hospital in Nepal.
2. To compare the pre and post training stress levels among participants of intervention and control group

Participants will Fill out the Depression, Anxiety and Stress Scale 21 and the Perceived Stress Scale before either being exposed to a 4-session stress management training (treatment group) or not being exposed to such training (control). All participants (both groups) will fill out the Depression, Anxiety and Stress Scale 21 and the Perceived Stress Scale for pre-post comparative measure.

DETAILED DESCRIPTION:
This study will aim to explore the effectiveness of a stress management program in nursing professionals in a community teaching hospital in Nepal. A 4-day stress management training program will be conducted and pre and post-training stress levels will be measured using the Perceived Stress Scale (PSS) and the Stress-Subscale of the Depression, Anxiety and Stress Scale-21 (DASS-21) one week prior to and after the training program. This experimental pre-post double arm study will involve 86 participants - all nursing staff from the Dhulikhel Hospital. Participants will be divided into 2 groups - treatment and control. The treatment group will be further divided into 2 groups of 20-25. The stress management training program will be held across 4 weeks with both groups receiving one training course each week (eg. Week 1 - session 1; Week 2 - session 2). Both questionnaires will be distributed again to both groups, 1 month after the last stress management session (1 - month follow up) .The control group whilst not being subjected to the Stress management training during the study period, will obtain the training upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* Nurses employed at the Dhulikhel Hospital
* Minimum one year work experience
* Minimum qualification certificate level of nursing
* Fluent in spoken and written English

Exclusion Criteria:

* Nurses with the post of nurse manager and above
* Nursing Students
* History having undergone stress management training in the past
* Absent for one or more sessions
* Incidence of a major stressful/critical life event during the study (e.g., divorce, death, and other critical events)

Ages: 8 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale - 21 | One week prior to 4-week intervention, one week and one month post-intervention.
  The DASS-21 is a 21-item tool measuring signs and symptoms of depression, anxiety and stress. The DASS-21 displays good to excellent internal consistency. Previous studies have reported a Cronbach's α ranging from 0.82 - 0.90 for Depression, .74 - .83 for Anxiety, and 82 - .87 for Stress. The DASS-21 has also been validated in Nepal with good reliability for each subscale, with Cronbach's alphas 0.79 for Anxiety, 0.91 for Stress, and 0.93 for Depression. Each item is on a 4-pint likert scale with higher scores indicating heightened symptoms of Depression, Anxiety and Stress.
Perceived Stress Scale | One week prior to 4-week intervention, one week and one month post-intervention.
  The PSS displays good internal consistency with a Cronbach's α ranging from 0.74 - 0.91. A Nepali version of the PSS has also been evaluated yielding validity, strong overall internal consistency (Cronbach's α = 0.95) and inter-rater reliability (ICC = 0.96). PSS scores can range from 0 to 56 with a higher score indicating higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Kavrepalanchowk, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behzadi S, Alizadeh Z, Samani NK, Ghasemi A, Fereidouni Z, Rostami K. Effect of stress management on job stress of intensive care unit nurses in hospitals affiliated to the University of Medical Sciences. Archivos Venezolanos de Farmacología y Terapéutica. 2021;40(8):824-7.
- [Background] Hakim RM, Walton LM, Schwartz JJ, Futrell SM, Zaaeed N, Raigangar VL. Nepali Version of the Ten-Item Perceived Stress Scale: Translation and Validation Study for Bhutanese Refugees. In2023 Combined Sections Meeting (CSM) 2023 Feb 25. APTA.
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Thapa DK, Visentin D, Kornhaber R, Cleary M. Psychometric properties of the Nepali language version of the Depression Anxiety Stress Scales (DASS-21). Nurs Open. 2022 Nov;9(6):2608-2617. doi: 10.1002/nop2.959. Epub 2021 Jun 23. PMID 34161668
- [Background] Zanon C, Brenner RE, Baptista MN, Vogel DL, Rubin M, Al-Darmaki FR, Goncalves M, Heath PJ, Liao HY, Mackenzie CS, Topkaya N, Wade NG, Zlati A. Examining the Dimensionality, Reliability, and Invariance of the Depression, Anxiety, and Stress Scale-21 (DASS-21) Across Eight Countries. Assessment. 2021 Sep;28(6):1531-1544. doi: 10.1177/1073191119887449. Epub 2020 Jan 9. PMID 31916468
- [Background] Pahlavanzadeh S, Asgari Z, Alimohammadi N. Effects of stress management program on the quality of nursing care and intensive care unit nurses. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):213-8. doi: 10.4103/1735-9066.180376. PMID 27186196
- [Background] Chaabane S, Chaabna K, Bhagat S, Abraham A, Doraiswamy S, Mamtani R, Cheema S. Perceived stress, stressors, and coping strategies among nursing students in the Middle East and North Africa: an overview of systematic reviews. Syst Rev. 2021 May 5;10(1):136. doi: 10.1186/s13643-021-01691-9. PMID 33952346
- [Background] Dutton S, Kozachik SL. Evaluating the Outcomes of a Web-Based Stress Management Program for Nurses and Nursing Assistants. Worldviews Evid Based Nurs. 2020 Feb;17(1):32-38. doi: 10.1111/wvn.12417. Epub 2020 Jan 8. PMID 31912984
- [Background] Mimura C, Griffiths P. The effectiveness of current approaches to workplace stress management in the nursing profession: an evidence based literature review. Occup Environ Med. 2003 Jan;60(1):10-5. doi: 10.1136/oem.60.1.10. PMID 12499451
- [Background] Ducharme F, Dubé V, Lévesque L, Saulnier D, Giroux F. An online stress management training program as a supportive nursing intervention for family caregivers of an elderly person. Canadian Journal of Nursing Informatics. 2011 Jun;6(2):1-9.
- [Background] Edwards D, Burnard P. A systematic review of stress and stress management interventions for mental health nurses. J Adv Nurs. 2003 Apr;42(2):169-200. doi: 10.1046/j.1365-2648.2003.02600.x. PMID 12670386
- [Background] Sailaxmi G, Lalitha K. Impact of a stress management program on stress perception of nurses working with psychiatric patients. Asian J Psychiatr. 2015 Apr;14:42-5. doi: 10.1016/j.ajp.2015.01.002. Epub 2015 Feb 7. PMID 25703040
- [Background] Lary A, Borimnejad L, Mardani-Hamooleh M. The Impact of a Stress Management Program on the Stress Response of Nurses in Neonatal Intensive Care Units: A Quasi-Experimental Study. J Perinat Neonatal Nurs. 2019 Apr/Jun;33(2):189-195. doi: 10.1097/JPN.0000000000000396. PMID 31021944
- [Background] Alkhawaldeh JMA, Soh KL, Mukhtar FBM, Peng OC, Anshasi HA. Stress management interventions for intensive and critical care nurses: A systematic review. Nurs Crit Care. 2020 Mar;25(2):84-92. doi: 10.1111/nicc.12489. Epub 2019 Dec 15. PMID 31840391
- [Background] Izdebski Z, Kozakiewicz A, Bialorudzki M, Dec-Pietrowska J, Mazur J. Occupational Burnout in Healthcare Workers, Stress and Other Symptoms of Work Overload during the COVID-19 Pandemic in Poland. Int J Environ Res Public Health. 2023 Jan 30;20(3):2428. doi: 10.3390/ijerph20032428. PMID 36767797
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Yazdani M, Rezaei S, Pahlavanzadeh S. The effectiveness of stress management training program on depression, anxiety and stress of the nursing students. Iran J Nurs Midwifery Res. 2010 Fall;15(4):208-15. PMID 22049282
- [Background] Pahlevani M, Ebrahimi M, Radmehr S, Amini F, Bahraminasab M, Yazdani M. Effectiveness of stress management training on the psychological well-being of the nurses. J Med Life. 2015;8(Spec Iss 4):313-318. PMID 28316750
- [Background] Kumar N, Jin Y. Impact of nurses' emotional labour on job stress and emotional exhaustion amid COVID-19: The role of instrumental support and coaching leadership as moderators. J Nurs Manag. 2022 Oct;30(7):2620-2632. doi: 10.1111/jonm.13818. Epub 2022 Oct 11. PMID 36181253
- [Background] Woo T, Ho R, Tang A, Tam W. Global prevalence of burnout symptoms among nurses: A systematic review and meta-analysis. J Psychiatr Res. 2020 Apr;123:9-20. doi: 10.1016/j.jpsychires.2019.12.015. Epub 2020 Jan 22. PMID 32007680
- [Background] Hersch RK, Cook RF, Deitz DK, Kaplan S, Hughes D, Friesen MA, Vezina M. Reducing nurses' stress: A randomized controlled trial of a web-based stress management program for nurses. Appl Nurs Res. 2016 Nov;32:18-25. doi: 10.1016/j.apnr.2016.04.003. Epub 2016 Apr 9. PMID 27969025